CLINICAL TRIAL: NCT02115932
Title: The Effectiveness of Strength and Balance Training in Patients With Diabetic Peripheral Neuropathy on Quality of Life and Functional Status: a Randomized Controlled Trial With Cost-utility Analysis
Brief Title: Effect of Physical Therapy in Improving the Health of Patients With Diabetic Peripheral Neuropathy
Acronym: DPN-QoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Kavita Venkataraman, Assistant Professor, Saw Swee Hock School of Public Health, National University of Singapore (NUS) and National University Health System (NUHS), National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NMRC/TA/0022/2013
Record Dates: First submitted 2014-04-11; First posted 2014-04-16 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Neuropathies; Peripheral Nervous System Diseases
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Complications; Diabetic Foot; Diabetic Neuropathies; Gait; Balance, Postural; Muscle Strength; Exercise Therapy; Physical Therapy Modalities; Endocrine System Diseases; Peripheral Nervous System Diseases; Metabolic Diseases; Glucose Metabolism Diseases; Quality of Life; Training
MeSH Terms: conditions — Diabetic Neuropathies; Peripheral Nervous System Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Complications; Diabetic Foot; Endocrine System Diseases; Metabolic Diseases | interventions — Exercise; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strength & Balance Training Intervention (Experimental): Subjects in this arm will undergo once weekly home-based strength and balance training for a period of 8 weeks.
  Interventions: Other: Strength & Balance Training
- Control (No Intervention): Subjects in this arm will not undertake any procedures or activities related to the study. They will continue with their prescribed medication and other medical advice from their treating physician as per usual.

INTERVENTIONS:
Other: Strength & Balance Training — Subjects will be guided through 8 weeks (1 hour per week) of home-based strength and balance training sessions. During each session, a trainer will guide subjects to perform muscle strengthening, range of motion, static balance, dynamic balance and endurance exercises, after an initial warm up. They will also be given advice on continuing such training as well as daily walking for the rest of the week.
  Other Names: Exercise Training; Gait Training; Motor Learning; Balance performance; Physical activity; Physiotherapy; Guided-exercise
  Arms: Strength & Balance Training Intervention

SUMMARY:
People with diabetes can have nerve damage in their extremities (peripheral neuropathy), and this can lead them to being less able to maintain their balance when they are standing, walking or performing complex movement tasks in their day-to-day life. This results in them being more prone to falls, and consequent injuries. The purpose of this study is to determine whether providing strength and balance retraining (in the form of specific physical exercises or activities) can help people with diabetic peripheral neuropathy regain their ability to maintain their balance, increase their confidence in performing balance-based activities and improve their quality of life.

DETAILED DESCRIPTION:
Individuals with diabetic peripheral neuropathy (DPN) comprise 16-24% of patients with diabetes mellitus in Singapore, and this is set to rise with the increasing prevalence of diabetes. DPN is also associated with the greatest reduction in health related quality of life (HRQoL) among all diabetic complications, specifically PCS (Physical health Component Summary) and its sub-components, physical functioning and physical role. However, there is currently no intervention that targets individuals with DPN for improvements in HRQoL and functional status.

The investigators hypothesise that a targeted intervention providing strength and balance training will improve HRQoL and functional status in patients with DPN, which will be sufficiently large relative to increases in cost to make the intervention cost-efficient.

The specific aims of the study are to test the effectiveness of a structured strength and balance training intervention in 1) improving the physical health component summary (PCS) measure of health related quality of life, 2) functional status, and 3) assessing cost-utility of the intervention, in individuals with diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 40 - 75
* Clinical diagnosis of Type II Diabetes Mellitus
* Presence of peripheral neuropathy (defined as neurothesiometer reading greater than 25 V and/or positive monofilament test in 2 or more sites in either foot)

Exclusion Criteria:

* Foot ulceration/ infection/ amputation
* Medical contraindication for physical activity or physiotherapy
* Non-diabetic neuropathy
* Orthopaedic/ Surgical/ Medical conditions affecting functional mobility and balance not due to diabetes or neuropathy (E.g. Stroke, Prosthesis use, Osteoarthritis)
* Retinopathy
* End-Stage Renal Disease requiring dialysis
* Congestive Heart Failure

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Change in Physical health component summary (PCS) of HRQoL from baseline at 2 and 6 months | Baseline, 2 and 6 months
  Physical Component Summary measured by SF-36 v2 questionnaire (norm-based score with mean of 50 and SD of 10 in general population)
Change in EQ5D HUI from baseline at 2 and 6 months | Baseline, 2 and 6 months
  Health Utility Index measured using EQ5D (range 0-1)

SECONDARY OUTCOMES:
Change in other domains of HRQoL from baseline at 2 and 6 months | Baseline, 2 and 6 months
  Domains of HRQoL measured by SF-36 v2 questionnaire ((norm-based score with mean of 50 and SD of 10 in general population)
Change in Functional Status from baseline at 2 and 6 months | Baseline, 2 and 6 months
  Functional Status measured using Timed Up and Go, Sit to Stand 5, Functional Reach, and activities based balance confidence tests
Change in static balance from baseline at 2 and 6 months | Baseline, 2 and 6 months
  static balance measured by a portable balance platform
Cost-utility of intervention measured by cost per Quality-Adjusted Life Year (QALY) gained | 2 months of intervention

OTHER OUTCOMES:
Change in muscle strength at ankle from baseline at 2 and 6 months | Baseline, 2 and 6 months
  muscle strength at ankle measured using a hand-held dynamometer
Change in range of motion at ankle and knee from baseline at 2 and 6 months | Baseline, 2 and 6 months
  range of motion at ankle and knee measured using a hand-held inclinometer
Number of subjects reporting falls and Injuries during the study | 6 months
  Subjected-reported falls and injuries
Change in gait from baseline at 2 and 6 months | Baseline, 2 and 6 months
  gait measured by a gait analysis platform

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Venkataraman, MBBS, PhD, Principal Investigator — National University of Singapore (NUS), and National University Health System (NUHS)
Locations (1):
- National University of Singapore; National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Venkataraman K, Wee HL, Leow MK, Tai ES, Lee J, Lim SC, Tavintharan S, Wong TY, Ma S, Heng D, Thumboo J. Associations between complications and health-related quality of life in individuals with diabetes. Clin Endocrinol (Oxf). 2013 Jun;78(6):865-73. doi: 10.1111/j.1365-2265.2012.04480.x. Epub 2013 Mar 25. PMID 22775311
- [Background] Alfonso-Rosa RM, Del Pozo-Cruz B, Del Pozo-Cruz J, Del Pozo-Cruz JT, Sanudo B. The relationship between nutritional status, functional capacity, and health-related quality of life in older adults with type 2 diabetes: a pilot explanatory study. J Nutr Health Aging. 2013 Apr;17(4):315-21. doi: 10.1007/s12603-013-0028-5. PMID 23538652
- [Background] Riandini T, Wee HL, Khoo EYH, Tai BC, Wang W, Koh GCH, Tai ES, Tavintharan S, Chandran K, Hwang SW, Venkataraman K. Functional status mediates the association between peripheral neuropathy and health-related quality of life in individuals with diabetes. Acta Diabetol. 2018 Feb;55(2):155-164. doi: 10.1007/s00592-017-1077-8. Epub 2017 Nov 28. PMID 29185052
- [Derived] Venkataraman K, Tai BC, Khoo EYH, Tavintharan S, Chandran K, Hwang SW, Phua MSLA, Wee HL, Koh GCH, Tai ES. Short-term strength and balance training does not improve quality of life but improves functional status in individuals with diabetic peripheral neuropathy: a randomised controlled trial. Diabetologia. 2019 Dec;62(12):2200-2210. doi: 10.1007/s00125-019-04979-7. Epub 2019 Aug 29. PMID 31468106